CLINICAL TRIAL: NCT03873714
Title: A Study of the Pipeline™ Vantage Embolization Device With Shield Technology™ for Endovascular Treatment of Wide-Necked Intracranial Aneurysms
Brief Title: Pipeline™ Vantage Embolization Device With Shield Technology™ for Wide-Necked Intracranial Aneurysms (ADVANCE)
Acronym: ADVANCE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study enrollment was halted on 14-Jun-2020. The study was not resumed and was terminated on 06-Jun-2024. Participants are no longer being examined or receiving intervention. Sponsor is no longer pursuing clinical evidence from the ADVANCE study.
Sponsor: Medtronic Neurovascular Clinical Affairs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COVSHLD0569
Record Dates: First submitted 2019-02-26; First posted 2019-03-13 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Pipeline™ Vantage Embolization Device with Shield Technology™ (Experimental): Pipeline™ Vantage Embolization Device with Shield Technology™
  Interventions: Device: Pipeline™ Vantage Embolization Device with Shield Technology™

INTERVENTIONS:
Device: Pipeline™ Vantage Embolization Device with Shield Technology™ — Pipeline™ Vantage Embolization Device with Shield Technology™
  Other Names: Pipeline™ Vantage

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of the Pipeline™ Vantage Embolization Device with Shield Technology™ in the treatment of intracranial aneurysms within the intended indication for use.

DETAILED DESCRIPTION:
The safety of the Pipeline™ Vantage will be assessed through incidence of major stroke in the territory supplied by the treated artery or neurological death at 1-year post-procedure. The effectiveness of the Pipeline™ Vantage will be assessed through incidence of complete aneurysm occlusion (Raymond Roy Scale Class 1) without significant parent artery stenosis (≤ 50%) or retreatment of the target aneurysm at 1-year post-procedure. Additional safety and effectiveness analyses will include incidence of major stroke in the territory supplied by the treated artery or neurological death at 2- and 3-years post-procedure, incidence of major stroke in the territory supplied by the treated artery or neurological death at 30 days post-procedure, incidence of delayed intraparenchymal hemorrhage >30 days post-procedure through 1-year post-procedure, incidence of subjects with disabling strokes that have a mRS decline to a score of 3 or more (mRS ≥ 3) due to a stroke-related cause assessed at a minimum of 90 days post-stroke event at 1 year, 2 year, and 3 year post-procedure, incidence of successful device implantation at the target site, incidence of complete aneurysm occlusion (Raymond Roy Class 1) at 1- and 3-years post-procedure, incidence of target aneurysm recurrence at 1- and 3-years post-procedure.

ELIGIBILITY:
Inclusion Criteria (Imaging):

* Subject has a target intracranial aneurysm located in the internal carotid artery (up to the terminus).
* Subject has a target intracranial aneurysm with an aneurysm neck ≥4mm or a dome-to-neck ratio of < 2.
* Subject has a target intracranial aneurysm that has a parent vessel with diameter 1.5-5.0 mm distal/proximal to the target intracranial aneurysm.

Inclusion Criteria (Clinical):

* Subject (or subject's legally authorized representative) has provided written informed consent using the IRB and Medtronic approved Informed Consent Form and agrees to comply with protocol requirements. HIPAA/data protection authorization has been provided and signed by the subject (or subject's legally authorized representative).
* Age 22-80 years at the time of consent.
* Life expectancy ≥3 years
* Subject has a mRS ≤ 2 at baseline to be determined by a certified independent assessor at the site.
* Subject has already been selected for endovascular treatment of the target aneurysm.
* Subject's last recorded P2Y12 reaction units (PRU) value is between ≥60 and ≤200 prior to study procedure.
* Subject has multiple increased risk factors for intracranial aneurysm rupture, including but not limited to, aneurysm morphology, smoking, hypertension, diabetes, age, prior and/or family history of rupture, and/or history of subarachnoid hemorrhage that may result in a benefit risk profile of endovascular treatment to outweigh the risks of intracranial aneurysm rupture during the subject's expected lifetime if left untreated.

Exclusion Criteria (Imaging):

* Subject has internal carotid artery bifurcation aneurysm.
* Aneurysms that arise from the Posterior Communicating Artery (PComm).
* The internal carotid artery aneurysms of the C7 segment will be excluded under the following conditions:

  1. Observed fetal posterior communicating artery (PComm) of fetal origin (A PComm of fetal origin is defined as a small, hypoplastic, or absent P1 segment of the posterior cerebral artery (PCA) with the PComm artery supplying a majority of blood flow to the P2 and higher order segments of the PCA)
  2. PComm overlapping with the aneurysm neck
  3. PComm branch arising from the dome of the aneurysm
* Subject has aneurysm arising from internal carotid artery but is primarily fed by posterior circulation (i.e., retrograde flow from the basilar artery) as confirmed by DSA

Exclusion Criteria (Clinical):

* Subject requires treatment of another aneurysm (with another treatment modality) within the affected territory of the target aneurysm during the study period.
* Subject has received an intracranial implant (e.g. coils) in the area of the target intracranial aneurysm within the past 6 months prior to the study procedure.
* Subject has had a SAH and/or target aneurysm rupture in the past 30 days prior to the study procedure.
* Subject has undergone a surgery including endovascular procedures in the last 30 days prior to the study procedure.
* Aneurysm vessel characteristics (e.g. parent vessel stenosis, irregular morphology) that would preclude the device from fully confirming to the parent vessel to reduce any risk of embolic complications, retreatment, or device movement.
* Subject has active vasospasm, malignant brain tumor or vascular malformation (e.g. arteriovascular malformation).
* History of major bleeding disorder (based on coagulation profile and platelet count) and/or subject presents with signs of active bleeding.
* Subject requires adjunctive device use (e.g. coils) during the index procedure.
* Subject has extradural target aneurysm <12mm which is not symptomatic or not exhibiting aneurysm growth (exception: unless it is a fusiform aneurysm <12 mm i.e., asymptomatic extradural fusiform aneurysms <12 mm can be included).
* Any known contraindication to treatment with the Pipeline™ Vantage Embolization Device with Shield Technology™, or use of antiplatelet therapy including:

  1. Active bacterial infection
  2. Contraindication to DAPT agents
* Pre-existing stent is in place in the parent artery at the target intracranial aneurysm location
* Platelet count < 100 x 10^3 cells/mm^3 or known platelet dysfunction.
* The Investigator determines that the health of the subject or the validity of the study outcomes (e.g., high risk of neurologic events, conditions that may increase the chance of stroke) may be compromised by the subject's enrollment.
* Subject is pregnant or wishes to become pregnant during the first year of study participation.
* Subject is participating in another clinical trial at any time during the duration of the study that could confound the treatment or outcomes of this investigation.
* Subject with known allergy to platinum or cobalt chromium alloy (including the major elements platinum, cobalt, chromium, nickel or molybdenum).
* History of previous acute ischemic stroke
* Subject is unable to undergo DSA or CTA imaging at follow-up

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2023-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Jabbour, MD, Principal Investigator — Thomas Jefferson University; Demetrius Lopes, MD, Principal Investigator — Advocate Health
Locations (3):
- United States (3):
  - Baptist Medical Center Jacksonville, Jacksonville, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - Stony Brook University Hospital, Stony Brook, New York

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be available.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was placed on an enrollment hold on 14 June 2020.
Pre-assignment Details: A total of 14 subjects were enrolled, of which seven (7) subjects were treated, six (6) subjects were withdrawn, and one (1) subject was a Screen Failure.
Groups:
- Study Group: Pipeline™ Vantage Embolization Device with Shield Technology™
Period: Overall Study
Arm/Group | Study Group
Started | 14
Primary Outcome Completion | 7
Completed | 7 (Six (6) were withdrawn, and one (1) was a Screen Failure.)
Not Completed | 7
Not completed — Six (6) were withdrawn, and one (1) was a Screen Failure | 7

BASELINE CHARACTERISTICS:
Arm/Group | Study Group
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (14.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Safety: Incidence of Major Stroke or Neurological Death
Description: Incidence of major stroke in the territory supplied by the treated artery or neurological death.
Time Frame: 1 year post-procedure
Population: All consented subjects in whom deployment of the Pipeline™ Vantage device was attempted
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 7
Participants | 1

2. Primary Outcome: Effectiveness: Incidence of Complete Aneurysm Occlusion
Description: Incidence of complete aneurysm occlusion (Raymond Roy Scale Class 1) without significant parent artery stenosis (≤ 50%) or retreatment of the target aneurysm at 1-year post-procedure.
Time Frame: 1 year post-procedure
Population: All consented subjects in whom deployment of the Pipeline™ Vantage device was attempted. Population data is inadequate for a complete primary effectiveness endpoint evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 7
Participants | 6

3. Secondary Outcome: Effectiveness: Incidence of Successful Device Implantation
Description: Incidence of successful device implantation at the target site
Time Frame: Day 0
Population: All Pipeline™ Vantage devices with deployment attempted
Measure: Count of Units; unit: Devices
Units Other Than Participants: Devices
Arm/Group | Study Group
Number analyzed (Participants) | 7
Number analyzed (Devices) | 10
Devices | 9

4. Secondary Outcome: Effectiveness: Incidence of Complete Aneurysm Occlusion
Description: Incidence of complete aneurysm occlusion (Raymond Roy Class 1)
Time Frame: 1 year post-procedure
Population: Subjects treated with Pipeline™ Vantage Embolization Device with Shield Technology™
Measure: Count of Participants; unit: Participants
Arm/Group | Pipeline™ Vantage Embolization Device With Shield Technology™
Number analyzed (Participants) | 7
Participants | 6

5. Secondary Outcome: Effectiveness: Incidence of Target Aneurysm Recurrence
Description: Incidence of target aneurysm recurrence at 1 year post-procedure
Time Frame: 1 year post-procedure
Population: Subjects treated with Pipeline™ Vantage Embolization Device with Shield Technology™
Measure: Count of Participants; unit: Participants
Arm/Group | Pipeline™ Vantage Embolization Device With Shield Technology™
Number analyzed (Participants) | 7
Participants | 0

6. Secondary Outcome: Safety: Incidence of Major Stroke
Description: Incidence of major stroke in the territory supplied by the treated artery or neurological death
Time Frame: 2 and 3 years post-procedure
Population: Subjects treated with Pipeline™ Vantage Embolization Device with Shield Technology™
Measure: Count of Participants; unit: Participants
Arm/Group | Pipeline™ Vantage Embolization Device With Shield Technology™
Number analyzed (Participants) | 7
Participants | 0

7. Secondary Outcome: Safety: Incidence of Major Stroke
Description: Incidence of major stroke in the territory supplied by the treated artery or neurological death
Time Frame: 30 days post-procedure
Population: All consented subjects in whom deployment of the Pipeline™ Vantage device was attempted.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 7
Participants | 1

8. Secondary Outcome: Safety: Incidence of Delayed Intraparenchymal Hemorrhage
Description: Incidence of delayed intraparenchymal hemorrhage >30 days post-procedure through 1-year post-procedure
Time Frame: >30 days post-procedure through 1 year post-procedure
Population: All consented subjects in whom deployment of the Pipeline™ Vantage device was attempted.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 7
Participants | 0

9. Secondary Outcome: Safety: Incidence of Subjects With Disabling Strokes
Description: Incidence of subjects with disabling strokes that have a mRS decline to a score of 3 or more (mRS ≥ 3) due to a stroke-related cause assessed at a minimum of 90 days post-stroke event
Time Frame: Assessed from procedure through 3 years post-procedure
Population: Subjects treated with Pipeline™ Vantage Embolization Device with Shield Technology™
Measure: Count of Participants; unit: Participants
Arm/Group | Pipeline™ Vantage Embolization Device With Shield Technology™
Number analyzed (Participants) | 7
Participants | 1

10. Secondary Outcome: Effectiveness: Incidence of Complete Aneurysm Occlusion
Description: Incidence of complete aneurysm occlusion (Raymond Roy Class 1)
Time Frame: 3 years post-procedure
Population: Subject that did not have complete occlusion at 1 year.
Measure: Count of Participants; unit: Participants
Groups:
- Pipeline™ Vantage Embolization Device With Shield Technology™: Subjects treated with Pipeline™ Vantage Embolization Device with Shield Technology™ that did not have complete occlusion at 3 years.
Arm/Group | Pipeline™ Vantage Embolization Device With Shield Technology™
Number analyzed (Participants) | 1
Participants | 0

11. Secondary Outcome: Effectiveness: Incidence of Target Aneurysm Recurrence
Description: Incidence of target aneurysm recurrence 3-years post-procedure
Time Frame: 3 years post-procedure
Population: Subjects treated with Pipeline™ Vantage Embolization Device with Shield Technology™
Measure: Count of Participants; unit: Participants
Groups:
- Pipeline™ Vantage Embolization Device With Shield Technology™: Subjects treated with Pipeline™ Vantage Embolization Device with Shield Technology™
Arm/Group | Pipeline™ Vantage Embolization Device With Shield Technology™
Number analyzed (Participants) | 6
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for each subject from the time of consent through 3 years post-procedure.
Description: Any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device. (ISO 14155:2011 3.2).
  MedDRA preferred term used for site reporting of adverse events.
Arm/Group | Study Group
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 2/7
Other Adverse Events (participants affected / at risk) | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=7)
Cerebral Hematoma (Nervous system disorders) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Cerebral Endovascular Aneurysm Repair (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=7)
Normocytic Anemia (Blood and lymphatic system disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Chest Pain (General disorders) | 1 (1)
Vascular Stent Stenosis (General disorders) | 1 (1)
Kidney Infection (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 2 (2)
Vascular Access Site Discharge (Injury, poisoning and procedural complications) | 1 (1)
Vascular Access Site Hematoma (Injury, poisoning and procedural complications) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Vaginal Hemorrhage (Reproductive system and breast disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cerebral Artery Stenosis (Nervous system disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Vasospasm (Vascular disorders) | 2 (4)
Constipation (Gastrointestinal disorders) | 1 (1) — Constipation
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was put on enrollment hold on 14 Jun 2020. At that time, fourteen (14) subjects had been enrolled and seven (7) subjects had been treated with the study device. All treated subjects were followed per protocol through the 3-year follow-up assessment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-02): https://cdn.clinicaltrials.gov/large-docs/14/NCT03873714/Prot_SAP_001.pdf